CLINICAL TRIAL: NCT00454012
Title: Use of Intrapartum Biophysical Profile When Fetal Heart Rate Monitoring is Non-reassuring in Labor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrolment
Sponsor: The Cooper Health System (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05046
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-03

CONDITIONS: Fetal Distress
Keywords: non reassuring fetal heart rate tracing; biophysical profile; assessing fetal wellbeing
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: biophysical profile

SUMMARY:
In this research project the investigators want to figure out whether ultrasound (a non-invasive method) can be used to assess how the fetus is doing during labor.

DETAILED DESCRIPTION:
When you are in labor, the heart beat of your fetus is monitored continuously. The normal pattern is reactive and suggests that the fetus is doing well. When the pattern is different from reactive, it is difficult to say if the fetus is doing well or not. Previous investigators have shown that even with the most worrisome fetal heart rate pattern, only 2/1000 cases would require immediate delivery. Currently, we use invasive procedures like taking a drop of blood from fetal head to further assess how the fetus is doing or just proceed with the fastest way of delivery (which could increase the risk associated with surgery). In this research project we want to figure out whether ultrasound (a non-invasive method) can be used to assess how the fetus is doing during labor.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous or induced labor
* Gestational ages between 35 - 42 weeks
* Singleton pregnancy
* Intrapartum non-reassuring or uninterpretable FHR tracing defined as any tracing that the Labor and Delivery obstetrician is uncomfortable about or feels does not absolutely provide fetal reassurance. Inclusive FHR patterns will be repetitive late decelerations, recurrent moderate to severe variable decelerations, reduced long or short-term variability, prolonged bradycardia (<120/min) that resolves, persistent fetal tachycardia (>160/min for >60 min,) or any other FHR patterns necessitating further fetal well being evaluation (like scalp pH or scalp stimulation).

Exclusion Criteria:

* Multiple gestation
* Gestational age < 35 weeks
* Patient denial to undergo ultrasound examination during labor
* Abnormal FHR tracing requiring stat delivery

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-04; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Meena Khandelwal, MD, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper UniversityHospital, Camden, New Jersey, United States

REFERENCES:
- [Result] Manning FA, Platt LD, Sipos L. Antepartum fetal evaluation: development of a fetal biophysical profile. Am J Obstet Gynecol. 1980 Mar 15;136(6):787-95. doi: 10.1016/0002-9378(80)90457-3. PMID 7355965